CLINICAL TRIAL: NCT01517581
Title: Study on the Association Between Brown Adipose Tissue Activation and White Adipose Tissue Accumulation in Successfully Treated Pediatric Malignancy
Brief Title: Brown Fat Activity and White Fat Accumulation
Status: Completed | Type: Observational
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Vicente Gilsanz, Professor, Children's Hospital Los Angeles
Other Study IDs: CHLA-Gilsanz-BAT/WAT
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Hodgkins Lymphoma; Non-hodgkins Lymphoma
Keywords: Brown adipose tissue
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Malignant Disease with no visualized BAT: Children 18 years or younger who 1) had PET/CT scans with evidence of malignant disease but no metabolically active brown adipose tissue (BAT) at diagnosis and 2) were disease free within 1 year of diagnosis.

SUMMARY:
White and brown adipocytes differ in their expression of hormones, cytokines, and inflammatory factors, and they modulate different biological functions. While white adipose tissue (WAT) serves as the primary site of energy storage, brown adipose tissue (BAT) instead metabolizes fat to produce heat and regulate body temperature. BAT is likely present in all humans, but the low prevalence of BAT depiction in adults and elderly subjects has hindered longitudinal assessments of the relation between BAT activity and WAT. Under typical imaging conditions, BAT is detected more frequently in children and teenagers than in adults with malignancy. Since most children with cancer have significantly shorter treatment courses and greater survival rates compared to adult patients, the investigators have the ability to examine the relation of repeated measures of body composition and BAT by selecting pediatric patients. In this study, the investigators will longitudinally examine whether BAT activity is related to changes in weight and the amounts of SAT, VAT, and abdominal muscle in children successfully treated for pediatric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients had PET/CT scans with evidence of malignant disease
* Patients had no metabolically active BAT at diagnosis on their PET/CT scan
* Patients were disease free within 1 year of diagnosis

Exclusion Criteria:

* Patients had PET/CT scans with no evidence of malignant disease
* Patients with metabolically active BAT at diagnosis on their PET/CT scan
* Patients were not disease free within 1 year of diagnosis

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with a history of malignancy such that they are required to undergo PET/CT exams.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2008-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Subcutaneous Adipose Tissue Volume at Follow-up | Baseline and up to 1 year
Change from Baseline in Visceral Adipose Tissue Volume at Follow-up | Baseline and up to 1 year
Change from Baseline in Presence of Brown Adipose Tissue | Baseline and up to 1 year
Change from Baseline in Abdominal Musculature Volume | Baseline and up to 1 year

SECONDARY OUTCOMES:
Change from Baseline in Anthropometric Measures at Follow-up | Baseline and up to 1 year
  Age, height, weight and BMI

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Gilsanz, MD, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Hamilton G, Smith DL Jr, Bydder M, Nayak KS, Hu HH. MR properties of brown and white adipose tissues. J Magn Reson Imaging. 2011 Aug;34(2):468-73. doi: 10.1002/jmri.22623. PMID 21780237
- [Result] Gilsanz V, Chung SA, Jackson H, Dorey FJ, Hu HH. Functional brown adipose tissue is related to muscle volume in children and adolescents. J Pediatr. 2011 May;158(5):722-6. doi: 10.1016/j.jpeds.2010.11.020. Epub 2010 Dec 18. PMID 21168855
- [Result] Gilsanz V, Smith ML, Goodarzian F, Kim M, Wren TA, Hu HH. Changes in brown adipose tissue in boys and girls during childhood and puberty. J Pediatr. 2012 Apr;160(4):604-609.e1. doi: 10.1016/j.jpeds.2011.09.035. Epub 2011 Nov 1. PMID 22048045
- [Result] Gilsanz V, Chung SA, Kaplowitz N. Differential effect of gender on hepatic fat. Pediatr Radiol. 2011 Sep;41(9):1146-53. doi: 10.1007/s00247-011-2021-7. Epub 2011 Mar 15. PMID 21404026
- [Result] Hu HH, Chung SA, Nayak KS, Jackson HA, Gilsanz V. Differential computed tomographic attenuation of metabolically active and inactive adipose tissues: preliminary findings. J Comput Assist Tomogr. 2011 Jan-Feb;35(1):65-71. doi: 10.1097/RCT.0b013e3181fc2150. PMID 21245691
- [Derived] Chalfant JS, Smith ML, Hu HH, Dorey FJ, Goodarzian F, Fu CH, Gilsanz V. Inverse association between brown adipose tissue activation and white adipose tissue accumulation in successfully treated pediatric malignancy. Am J Clin Nutr. 2012 May;95(5):1144-9. doi: 10.3945/ajcn.111.030650. Epub 2012 Mar 28. PMID 22456659